CLINICAL TRIAL: NCT02966184
Title: Comparison of Benzalkonium Chloride Containing Albuterol Versus Preservative Free Albuterol for the Treatment of Status Asthmaticus
Brief Title: Comparison of Albuterol for Status Asthmaticus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study Drug Backorder
Sponsor: Norton Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16.0721
Record Dates: First submitted 2016-10-26; First posted 2016-11-17 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Status Asthmaticus
MeSH Terms: conditions — Status Asthmaticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benzalkonium chloride (BAC) Albuterol (No Intervention): This arm includes the current standard of care which patients receive at the institution. No interventions will be made within this group of patients.
- Preservative Free Albuterol (Experimental): This arm includes the preservative free albuterol which is being investigated. Treatment for this arm will follow current standards of care, with the only difference being the albuterol formulation.
  Interventions: Drug: preservative free albuterol

INTERVENTIONS:
Drug: preservative free albuterol — Preservative free albuterol for nebulization
  Other Names: Albuterol Sulfate Inhalation Solution 0.5%; 0487-9901-02; 0487-9901-30
  Arms: Preservative Free Albuterol

SUMMARY:
This study is designed to compare the length of continuous albuterol administration between two different albuterol formulations, BAC containing albuterol versus preservative free albuterol.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the length of continuous albuterol administration between patients receiving BAC containing albuterol versus preservative free albuterol. Secondary objectives include comparison of therapy escalation, asthma scores, forced expiratory volume in one second (FEV1) at discharge, length of hospital stay, and cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study if they are admitted to the 5th floor of Norton Children's Hospital for the treatment of an acute asthma exacerbation, initiated on continuous albuterol inhalation therapy, and are between 5 and 17 years of age.

Exclusion Criteria:

* Patients will be excluded from the study if they are transferred from the 5th floor to the Pediatric Intensive Care Unit (PICU), admitted for any indication other than acute asthma exacerbation, or removed from the inpatient asthma protocol for any given reason.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Murray, PharmD, Principal Investigator — Norton Healthcare
Locations (1):
- Norton Children's Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made sharable.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: According to the study design, we had to assent/consent (but not enrolled) far more patients than would be eligible for study inclusion/enrollment. This was to prevent a delay in therapy if the patient needed to be administered continuous albuterol immediately. Most consented patients did not get assigned to one of the 'study nursing units' so they were not eligible for study enrollment. Only 8 patients met the criteria for enrollment.
Groups:
- Benzalkonium Chloride-Containing Albuterol: This arm includes the current standard of care (preservative-containing albuterol nebulization) which patients receive at the institution. No interventions will be made within this group of patients.
- Preservative-Free Albuterol: This arm includes the preservative-free albuterol nebulization which is being investigated. Treatment for this arm will follow current standards of care, with the only difference being the albuterol formulation.
Period: Overall Study
Arm/Group | Benzalkonium Chloride-Containing Albuterol | Preservative-Free Albuterol
Started | 0 | 8
Completed | 0 | 0
Not Completed | 0 | 8

BASELINE CHARACTERISTICS:
Population: There were no patients enrolled in the Benzalkonium Chloride-Containing Albuterol group
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzalkonium Chloride-Containing Albuterol | Preservative-Free Albuterol | Total
Number analyzed (Participants) | 0 | 8 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 7.78 (2.46) | 7.78 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 3
  Male |  | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 6 | 6
  White |  | 2 | 2
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Albuterol Administration
Description: Length of continuous albuterol administration between patients receiving BAC containing albuterol versus preservative free albuterol during hospital admission for status asthmaticus
Time Frame: Hours until discontinuation of therapy, an average of 72 hours
Population: Study was terminated due to medication backorder and therefore outcome data collection was never performed nor analyzed
Arm/Group | Benzalkonium Chloride-Containing Albuterol | Preservative-Free Albuterol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected only during the patient's admission. Follow-up assessment after discharge did not occur
Description: Our definition of adverse event and or serious adverse event did not differ from clinicaltrials.gov
Arm/Group | Benzalkonium Chloride-Containing Albuterol | Preservative-Free Albuterol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/8
Other Adverse Events (participants affected / at risk) | 0/0 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02966184/Prot_SAP_000.pdf